CLINICAL TRIAL: NCT06145841
Title: Clinical Application of Metagenomic Next-Generation Sequencing-Guided Anti-Infection Strategies in AIDS Patients With Severe Pneumonia and/or Sepsis
Brief Title: Metagenomic Next-Generation Sequencing Guides Anti-Infection Strategies
Status: Recruiting | Type: Observational
Sponsor: Guangzhou 8th People's Hospital (Other)
Responsible Party: Principal Investigator, Linghua LI, Chief physician, Guangzhou 8th People's Hospital
Other Study IDs: GZ8H-202322259s
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: AIDS; Pneumonia; Sepsis, Neonatal
Keywords: AIDS; severe pneumonia; Sepsis; metagenomic next-generation sequencing
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Pneumonia; Neonatal Sepsis; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Reserved biological samples are derived from peripheral blood specimens, used for pathogen metagenomic next-generation sequencing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pathogen metagenomic next-generation sequencing group: This group uses metagenomic next-generation sequencing along with traditional pathogen detection techniques to test for infectious pathogens. The follow-up times are the 1st, 2nd, 3rd, and 4th weeks after being diagnosed with severe pneumonia or sepsis.
  Interventions: Diagnostic Test: Pathogen metagenomic next-generation sequencing
- Conventional pathogen detection group: This group only used conventional pathogen detection methods for the identification of infectious pathogens. Follow-up was conducted at the 1st, 2nd, 3rd, and 4th weeks after the diagnosis of severe pneumonia or sepsis. The conventional means of pathogen detection include, but are not limited to, fungal serology tests, cryptococcal capsular antigen detection, CMV-DNA tests, sputum smear microscopy, gamma interferon release assays, Xpert MTB/RIF, BLAF culture, blood and bone marrow cultures, radiological examinations, and histopathological examinations.

INTERVENTIONS:
Diagnostic Test: Pathogen metagenomic next-generation sequencing — In diagnosing patients with AIDS combined with severe pneumonia and/or sepsis, use pathogen metagenomics technology to detect peripheral blood specimens
  Groups: Pathogen metagenomic next-generation sequencing group

SUMMARY:
This study aims to observe the effectiveness of clinical application in guiding anti-infection treatments in AIDS patients with severe pneumonia and/or sepsis using Metagenomic Next-Generation Sequencing-based technology in the real world

DETAILED DESCRIPTION:
The study focuses on AIDS patients with severe pneumonia and/or sepsis, divided into groups based on whether metagenomic next-generation sequencing technology is used in the real world or not. The groups are the metagenomic next-generation sequencing group and the conventional pathogen detection group, with metagenomic sequencing samples derived from blood specimens. The study compares the pathogen detection rates and clinical diagnosis conformity rates of the aforementioned groups, as well as the efficiency of diagnosis in guiding clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV infection;
2. Progression to AIDS stage: CD4+ count <200 cells/ul and/or occurrence of AIDS opportunistic infections;
3. Age between 18 and 65 years;
4. Meeting the diagnosis of severe pneumonia or septic shock:

   1. The criteria for severe pneumonia diagnosis refer to the 2021 ATS (American Thoracic Society) and IDSA (Infectious Diseases Society of America) guidelines for the treatment of community-acquired pneumonia;
   2. The criteria for septic shock refer to the Chinese Society of Critical Care Medicine's "Chinese Guidelines for the Emergency Treatment of Sepsis/Septic Shock (2018).

Exclusion Criteria:

1. Coexisting central nervous system lesions, severe liver disease, or cirrhosis;
2. Concurrent AIDS-related or unrelated tumors;
3. Women who are pregnant or breastfeeding;
4. Severe underlying diseases of the heart, lungs, liver, kidneys, etc.;
5. Alcohol abuse or drug use;
6. The researcher believes that the overall condition of the subject affects the evaluation and completion of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study participants come from the OSPWH (Patients With HIV/AIDS) cohort at the Guangzhou Eighth People's Hospital.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2026-10-23 (Estimated); Study Completion 2027-10-23 (Estimated)

PRIMARY OUTCOMES:
Pathogen detection rate and clinical diagnosis concordance rate | 4 weeks
  Analyze the concordance rate between the pathogen spectrum detected using pathogen metagenomics technology and the final clinical disease diagnosis.

SECONDARY OUTCOMES:
Clinical treatment efficacy rate | 4 weeks
  "Clinical treatment efficacy includes: 1) AIDS combined with severe pneumonia: pathogen clearance or quantitative change, PSI score, chest X-ray/chest CT; 2) AIDS combined with sepsis: pathogen clearance or quantitative change, SOFA score.

CONTACTS AND LOCATIONS:
Locations (1):
- Linghua Li, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barbier F, Mer M, Szychowiak P, Miller RF, Mariotte E, Galicier L, Bouadma L, Tattevin P, Azoulay E. Management of HIV-infected patients in the intensive care unit. Intensive Care Med. 2020 Feb;46(2):329-342. doi: 10.1007/s00134-020-05945-3. Epub 2020 Feb 3. PMID 32016535
- [Result] Besser J, Carleton HA, Gerner-Smidt P, Lindsey RL, Trees E. Next-generation sequencing technologies and their application to the study and control of bacterial infections. Clin Microbiol Infect. 2018 Apr;24(4):335-341. doi: 10.1016/j.cmi.2017.10.013. Epub 2017 Oct 23. PMID 29074157
- [Result] Pei F, Yao RQ, Ren C, Bahrami S, Billiar TR, Chaudry IH, Chen DC, Chen XL, Cui N, Fang XM, Kang Y, Li WQ, Li WX, Liang HP, Lin HY, Liu KX, Lu B, Lu ZQ, Maegele M, Peng TQ, Shang Y, Su L, Sun BW, Wang CS, Wang J, Wang JH, Wang P, Xie JF, Xie LX, Zhang LN, Zingarelli B, Guan XD, Wu JF, Yao YM; Shock and Sepsis Society of Chinese Research Hospital Association; China Critical Care Immunotherapy Research Group; International Federation of the Shock Societies (IFSS). Expert consensus on the monitoring and treatment of sepsis-induced immunosuppression. Mil Med Res. 2022 Dec 26;9(1):74. doi: 10.1186/s40779-022-00430-y. PMID 36567402